CLINICAL TRIAL: NCT04422067
Title: Usefulness of Cephalometry in the Second and Third Trimester of Pregnancy in the Diagnosis of Fetal Microretrognathia : Prenatal Cephal
Brief Title: Usefulness of Cephalometry in the Second and Third Trimester of Pregnancy in the Diagnosis of Fetal Microretrognathia
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0295
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Pierre Robin Sequence
Keywords: with one or more fetuses suffering from a microretrognathia; Cephalometry; Prenatal Diagnosis; Facial angles; Fetal echography; Microretrognathia; diagnosed prenatally
MeSH Terms: conditions — Pierre Robin Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group (Retrognatism): All pregnant patients with one or more fetuses suffering from a microretrognathia, diagnosed prenatally and integrated into a Pierre Robin Sequence, were included. All cases were confirmed postnatally, either by a pediatric examination or by a fetopathological examination in the case of a medical termination of the pregnancy. We had 21 cases.
  Interventions: Other: Fetal cephalometry
- Control group: 47 pregnant patients with fetus without facial abnormalities
  Interventions: Other: Fetal cephalometry

INTERVENTIONS:
Other: Fetal cephalometry — Fetal cephalometry

SUMMARY:
Congenital retrognathia, with or without Pierre Robin Sequence (PRS), is a rare anomaly which can be associated with chromosomal abnormalities. Respiratory and feeding consequences can be present at birth. After birth, the diagnosis of retrognathia is based on the clinical examination. Cephalometry can be used to complete the diagnosis. Several authors have proposed the use of objective quantitative ultrasound parameters for the antenatal screening of PRS. In our study, the investigators evaluated fetal cephalometry.

The aim First, the investigators studied the inter- and intra-observer reproducibility of cephalometry. Second, the investigators established reference values for antenatal cephalometry in normal fetuses. Third, the investigators compared the diagnostic performance of cephalometry and the other angles described in the literature for the diagnosis of retrognathia.

ELIGIBILITY:
Inclusion criteria:

* Pregnant patient (Aged >18years old)
* with one or more fetuses suffering from a microretrognathia
* diagnosed prenatally
* integrated into a Pierre Robin Sequence

Exclusion criteria:

* Uncvertain diagnosis
* Absence of 3D rendering volume

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All pregnant patients with one or more fetuses suffering from a microretrognathia, diagnosed prenatally and integrated into a Pierre Robin Sequence
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Reproducibility of cephalometry | During ultrasound
  Reproducibility of cephalometry

SECONDARY OUTCOMES:
Perfomance of several angle to diagnose retrognatism | During ultrasound
  Perfomance of several angle to diagnose retrognatism

CONTACTS AND LOCATIONS:
Overall Officials: Florent FUCHS, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC